CLINICAL TRIAL: NCT01199159
Title: A Pilot Study of the Preoperative Misoprostol in Reducing Operative Blood Loss During Hysterectomy
Brief Title: Preoperative Misoprostol in Reducing Blood Loss in Total Abdominal Hysterectomy (TAH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Joyce Chai, University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: misohys001
Record Dates: First submitted 2010-09-06; First posted 2010-09-10 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-09

CONDITIONS: Hysterectomy
Keywords: misoprostol; hysterectomy; operative blood loss; total abdominal hysterectomy
MeSH Terms: interventions — Misoprostol; Vitamin B 6

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- preoperative misoprostol (Active Comparator): 400mcg misoprostol given preoperatively
  Interventions: Drug: Misoprostol
- Placebo (Placebo Comparator)
  Interventions: Drug: Vitamin B 6

INTERVENTIONS:
Drug: Misoprostol — 400mcg misoprostol given sublingually 30 minutes before total abdominal hysterectomy
  Arms: preoperative misoprostol
Drug: Vitamin B 6 — 20mg vitamin B6 given sublingually 30 minutes before total abdominal hysterectomy
  Arms: Placebo

SUMMARY:
Total abdominal hysterectomy is known to be associated with operative blood loss, which can lead to patients' morbidity. Misoprostol, a prostaglandin, has been shown to be effective in reducing operative blood loss during myomectomy. It is the first study to investigate if preoperative misoprostol is effective in reducing operative blood loss during total abdominal hysterectomy.

DETAILED DESCRIPTION:
Uterine leiomyoma is the commonest benign tumour affecting women in their reproductive age. Around 20-50% can cause symptoms that warrant treatment. Different medical therapies, including gonadotrophin releasing hormone analogues, mifepristone, progestins and androgens have been tried. However, most of the medical therapy have significant side-effects that would only allow a short-term treatment. Total abdominal hysterectomy is the definitive treatment for large, symptomatic fibroids. Operative mortality of total abdominal hysterectomy is rare. However, the operation may be associated with significant morbidities. Significant operative blood loss that required blood transfusion and oral iron supplement is not uncommonly encountered after total abdominal hysterectomy.

Various methods have been tried to reduce the operative blood loss during total abdominal hysterectomy. A course of hormonal therapy for a few months before operation aiming to shrink the size of fibroid(s) and reduce the vascularity is the commonest approach. Although it is effective, there are significant side effects and the cost of gonadotrophin releasing hormone analogues is high. Intramyometrial vasopressin injection has been reported, but serious complications have been reported.

Misoprostol, a prostaglandin E1 analogue, has been widely used in clinical practice in obstetrics and gynaecology. It stimulates uterine contractions and this increase in myometrial contraction will lead to contraction of the vessels supplying blood to the leiomyomas. Misoprostol has also been shown to increase the uterine artery resistance and reduce the blood flow to the leiomyomas. Study by Celik et al has shown that pre-operative misoprostol can reduce intra-operative blood loss and need for post-operative blood transfusion after abdominal myomectomy. Chang et al investigated the use of misoprostol and oxytocin in laparoscopy-assisted vaginal hysterectomy and found that the combination of pre-operative misoprostol and intra-operative oxytocin can reduce blood loss by 200 ml. As misoprostol can stimulate uterine contraction and reduce uterine blood flow, based on the hypothesis that pre-operative misoprostol may redistribute the blood from the diseased uterus back to the circulation hence reducing operative blood loss during total abdominal hysterectomy, we use a double-blind randomized controlled trial to investigate whether a single dose of sublingual misoprostol before total abdominal hysterectomy +/- salpingo-oophorectomy for symptomatic uterine leiomyomas can reduce operative blood loss and need for post-operative blood transfusion.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic women undergoing total abdominal hysterectomy for various benign gynaecological diseases in Queen Mary Hospital

Exclusion Criteria:

* any contraindication to misoprostol, including mitral stenosis, glaucoma, sickle cell anaemia, diastolic pressure over 100mmHg, severe asthma, or known allergy to prostaglandin;
* a known history of pelvic/ovarian endometriosis;
* a known history of or active medical disease;
* a known history of previous myomectomy;
* women who had pre-operative mifepristone or gonadotrophin releasing hormone analogues treatment;
* women with mental impairment or incompetent in giving consent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2007-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
operative blood loss | duration of operation, up to 3 hours
  The total volume of blood loss was estimated by measuring the amount of blood accumulated in the aspiration equipment and the amount of blood on the surgical gauze using a alkaline haematin method.

SECONDARY OUTCOMES:
the requirement of blood transfusion | from intra-operation to hospital discharge, up to 7 days
the change in haemoglobin level after operation | preoperative to 30 hours postoperative
the incidence of side effects | 30 minutes after misoprostol/placebo was given

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Chai J, Hon E, Li CF, Pun TC, Yeung SB, Ho PC. A pilot study of pre-operative misoprostol in reducing operative blood loss during hysterectomy. Eur J Obstet Gynecol Reprod Biol. 2011 Sep;158(1):72-5. doi: 10.1016/j.ejogrb.2011.03.023. Epub 2011 Apr 23. PMID 21514988